CLINICAL TRIAL: NCT05506072
Title: Blood Flow Restriction Training Versus Standard Physical Therapy After Shoulder Stabilization Surgery: A Randomized Controlled Trial.
Brief Title: Blood Flow Restriction Training Versus Standard Physical Therapy After Shoulder Stabilization Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamie Morris, Director and Professor, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KACH.2022.0058; 22KACH005 (Other: Keller)
Record Dates: First submitted 2022-08-10; First posted 2022-08-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anterior Shoulder Dislocation; Recurrent Shoulder Dislocation; Shoulder Subluxation; Surgery
MeSH Terms: conditions — Shoulder Dislocation | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BFR group with standard therapy (Experimental): Participants will be randomized into their assigned group of receiving standard therapy with BFR by a blinded therapist within the study. Participants will then visit the clinic for study testing at six weeks, 12 weeks, and six months after their surgery. During each of these visits, they will be asked to complete a survey, and then their shoulder strength and flexibility will be measured. Each study visit will last approximately 30 minutes. Participants will also attend 12-18 shoulder rehabilitation sessions in the clinic over six weeks from the six week to 12 week mark (about two to three sessions per week). Each rehabilitation session will last approximately 30 minutes and consist of Blood Flow Restriction Training with the standard rehabilitation exercises. Between the 12-week follow-up and 6-month follow-up, participants will receive standard post-surgical rehabilitation for their specific shoulder surgery without Blood Flow Restriction training.
  Interventions: Other: Blood flow restriction therapy; Other: Standard Physical Thearapy
- standard therapy group (Active Comparator): Participants will be randomized into their assigned group of receiving standard therapy without BFR by a blinded therapist within the study using a computer generated randomization formula Participants will then visit the clinic for study testing at six weeks, 12 weeks, and six months after their surgery. During each of these visits, they will be asked to complete a survey, and then their shoulder strength and flexibility will be measured. Each study visit will last approximately 30 minutes. Participants will also attend 12-18 shoulder rehabilitation sessions in the clinic over six weeks from the six week to 12 week mark (about two to three sessions per week). Each rehabilitation session will last approximately 30 minutes and consist of standard rehabilitation exercises without BFR.
  Between the 12-week follow-up and 6-month follow-up, participants will receive standard post-surgical rehabilitation for their specific shoulder surgery without Blood Flow Restriction training.
  Interventions: Other: Blood flow restriction therapy

INTERVENTIONS:
Other: Blood flow restriction therapy — Blood Flow Restriction involves the application of a tourniquet to an extremity to partially restrict the arterial and venous blood flow to stimulate localized cellular and systemic hormonal changes that occur in high intensity exercise. BFR Training may produce similar cellular and muscular responses to cause hypertrophy when exercise is performed at low intensity. Studies have compared BFR therapy in the lower extremities with light load resistance exercise to light load resistance alone and observed greater improvements in the BFR group. A recent systematic review further identified that adding BFR to exercise effectively augments muscle strength and size. Additionally, BFR has been shown to be applied in a safe manner with low risk for complications. With this growing body of evidence supporting BFR, it is becoming increasingly common in rehabilitation
Other: Standard Physical Thearapy — Participants will be randomized into their assigned group of receiving standard therapy without BFR by a blinded therapist within the study using a computer generated randomization formula Participants will then visit the clinic for study testing at six weeks, 12 weeks, and six months after their surgery. During each of these visits, they will be asked to complete a survey, and then their shoulder strength and flexibility will be measured. Each study visit will last approximately 30 minutes. Participants will also attend 12-18 shoulder rehabilitation sessions in the clinic over six weeks from the six week to 12 week mark (about two to three sessions per week). Each rehabilitation session will last approximately 30 minutes and consist of standard rehabilitation exercises without BFR.
  Between the 12-week follow-up and 6-month follow-up, participants will receive standard post-surgical rehabilitation for their specific shoulder surgery without Blood Flow Restriction training.
  Arms: BFR group with standard therapy

SUMMARY:
Describe the purpose and objective(s) of the study, specific aims, and/or research questions/hypotheses:

The purpose of this Randomized Controlled Trial is to evaluate the effectiveness of Blood Flow Restriction (BFR) training with standard care of physical therapy versus the standard care of Physical Therapy alone and its effect on shoulder function and patient outcomes in military cadets recovering from shoulder stabilization surgery. We hypothesize after 6 weeks of BFR training will contribute to 13 (76%) or more participants will achieve scores within one standard deviation of normative values for isometric strength and functional tests at six months following shoulder stabilization surgery.

Furthermore, we hypothesize that 14 (82%) or more participants will report improved patientreported outcomes as determined by the minimal clinical difference (MCD) at 12 weeks and six months post-operatively. Objective 1: To evaluate the effectiveness of blood flow restriction (BFR) training on shoulder isometric strength, as measured by a digital handheld dynamotor following shoulder stabilization surgery in military cadets. Objective 2: To evaluate the effectiveness of blood flow restriction (BFR) training on shoulder range of motion, as measured by a digital inclinometer, following shoulder stabilization surgery in military cadets. Objective 3: To evaluate the effectiveness of blood flow restriction (BFR) training on shoulder function as measured by the Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST), Seated Shot-Put Test (SSPT), and Upper Quarter Y-Balance Test (UQYBT), following shoulder stabilization surgery in military cadets. Objective 4: To evaluate the effectiveness of BFR training on shoulder pain, measured by a numerical pain rating scale, following shoulder stabilization surgery in military cadets.

Objective 5: To evaluate the effectiveness of a BFR training on patient-reported outcomes, measured by Single Assessment Numeric Evaluation (SANE), Shoulder Pain and Disability Index (SPADI), and the Quick Disabilities of Arm, Shoulder and Hand (DASH) following shoulder stabilization surgery in military cadets. Aim 1:To identify whether BFR with Physical Therapy is more effective at increasing shoulder strength than therapy alone following shoulder stabilization surgery. We hypothesize that the BFR with Physical Therapy group will be more effective at increasing shoulder strength than the Physical Therapy group without BFR following shoulder stabilization surgery. Aim 2:To identify whether BFR with Physical Therapy is more effective at increasing shoulder function than therapy alone following shoulder stabilization surgery. We hypothesize that the BFR with Physical Therapy group will be more effective at increasing shoulder function than the Physical Therapy group without BFR following shoulder stabilization surgery.

DETAILED DESCRIPTION:
During study:

Participants will be recruited from the Keller Army Community Hospital (KACH) the KACH Orthopedic Clinic and the Arvin Cadet Physical Therapy Clinic. Participants will be screened for possible benefits of participation and related inclusion

/exclusion criteria as is done within traditional means by the referring provider.

Participant recruitment and briefing by the lead primary investigator (PI) or associate investigator (AI) will be conducted.

Participants wishing to participate in the study will undergo informed consent process with PI or AI. Participants agreeing to participate will complete consent by signing an informed consent form and HIPAA authorization form. All data will be recorded and stored by the subject identification number. Participants will be randomized into their assigned group of either receiving standard therapy with Blood Flow Restriction (BFR) or standard therapy alone by a blinded therapist within the study using a computer generated randomization formula Participants will then visit the clinic for study testing at six weeks, 12 weeks, and six months after their surgery. During each of these visits, they will be asked to complete a survey, and then their shoulder strength and flexibility will be measured. Each study visit will last approximately 30 minutes. Participants will also attend 12-18 shoulder rehabilitation sessions in the clinic over six weeks from the six week to 12 week mark (about two to three sessions per week). Each rehabilitation session will last approximately 30 minutes and consist of Blood Flow Restriction Training and/or standard rehabilitation exercises. Between the 12-week follow-up and 6-month follow-up, participants will receive standard post-surgical rehabilitation for their specific shoulder surgery without Blood Flow Restriction training. Baseline Testing All participants will undergo baseline testing at 6 weeks in the following order: 1.

Demographic data 2. self-report outcome measures; 3. Range of motion (ROM) testing; 4.

isometric strength testing. Initial patient reported outcome measures will be recorded on the Numerical Pain Rating Scale (NPRS), the Single Assessment Numeric Evaluation (SANE), the Shoulder Pain and Disability Index (SPADI), and the Quick Disabilities of Arm, Shoulder, Hand (DASH).

Initial shoulder flexion, external rotation (ER), and internal rotation (IR) Range of Motion (ROM) measurements will be conducted using the digital inclinometer Initial shoulder isometric abduction, ER, and IR strength will be assessed using a handheld dynamometer. Intervention Participants will either receive the current standard of care in post-operative shoulder stabilization rehabilitation without BFR training during each treatment session or current standard of care in post-operative shoulder stabilization rehabilitation plus BFR training.

BFR will be done via Delfi Portable Tourniquet System (BFR (Delfi Medical Innovations Inc., Vancouver, Canada) All participants will perform their rehabilitation a minimum of two times per week in the rehabilitation clinic. Patient contact time with their medical providers will be the same in both groups. The BFR treatment with the BFR group will be applied during each treatment session for 6 weeks (weeks 6-12). Pain will be assessed at the beginning and end of each treatment session using the Numerical Pain Rating Scale, in accordance with standard clinical practice. Exercise intensity will be determined each session using the OMNI res scale and participants will use that load for their daily exercises. The BFR group will exercise at an intensity of 2-3 on the OMNI res scale on the involved side and then exercise at a 6-8 on the uninvolved side. The non-BFR group will exercise at a 6-8 on the involved and uninvolved side. These loads will be annotated and used be referred to when completing strengthening exercises. Participants will then perform a 30-minute session of rehabilitation. The BFR group will apply the BFR tourniquet and it will be inflated to 50% Limb Occlusion Pressure (LOP) throughout the duration of the treatment. The upper body aerobic exercise will be performed on an upper body cycle (UBC). Intensity will be determined by the perceived exertion of OMNI Res at a resistance the participant considers easy(2-3). The strengthening exercises will consist of three unilateral standing exercises to be performed on both upper extremities. The exercises to be performed are ER with the shoulder adducted to the thorax, scapular retraction with a combined low row, and flexion in scapular plane. Each exercise will be performed while standing using Keiser Functional Trainer (Keiser Corp model 003025.15, Fresno, CA). The resistance for the strengthening exercises will be selected as described above using the Omni res scale. All participants will perform 75 repetitions in total per exercise broken in to 4 sets (30,15,15,15). A 30 second rest period will be issued between exercises. Participants will be permitted to increase or decrease the resistance as needed to stay within the specified perceived exertion range but will be annotated for any deviation from pre-load assessment. The treatment session will end when a participant completes all sets and repetitions for each exercise. However, if a participant is unable to complete all exercises in 30 minutes, the BFR cuff will be deflated and removed. Then, the participant will finish the exercises without BFR. Patients will also perform a home exercise program(HEP) that reinforces the in-clinic treatment. Compliance with the home exercise program will be documented by a patient log to be completed daily and turned into the project manager weekly. All groups will perform their HEP strength exercises at same perceived load intensity of a 6-8 on the OMNI res scale. Assessments (6 weeks); Follow up (12-week, and 6 months post-surgery)

All participants will undergo baseline and follow-up testing in the following order: 1. self report outcome measures; 2. Range of motion testing; 3. isometric strength testing; 4. Functional testing at 6-month follow-up only Follow-up patient reported outcome measures will be recorded on the Numerical Pain Rating Scale (NPRS), the Single Assessment Numeric Evaluation (SANE), the Shoulder Pain and Disability Index (SPADI), and the Quick Disabilities of Arm, Shoulder, Hand (DASH). Shoulder flexion, external rotation (ER), and internal rotation (IR) Range of Motion (ROM) measurements will be conducted using the digital inclinometer Shoulder isometric abduction, ER, and IR strength will be assessed using a hand-held dynamometer. Functional tests will be conducted in the same order: Closed Kinetic Chain Upper Extremity Stability Test (CKQUEST), Upper Quarter Y Balance Test (UQYBT), Seated Shotput Test (SSPT) Study participation completed after the 6-month follow-up

ELIGIBILITY:
Inclusion Criteria:

1. enrolled in the US Military Academy as a Cadet?
2. between the age of 17 to 30 years?
3. USMA cadet who was diagnosed with unilateral or multi-directional instability who underwent primary or revised surgery as well as open and arthroscopic shoulder stabilization surgery procedures at KACH.
4. near 6 weeks post-operative at start and will be cleared to begin strengthening exercises at that time

Exclusion Criteria:

1. Have not had a rotator cuff surgery with the current surgical repair?
2. Have not had a humeral neck or shaft fracture?
3. Had not had a history of head, neck, or shoulder procedures requiring general anesthesia within 6 weeks from surgery
4. Have not had a history of deep vein thrombosis (DVT) within the 12 months from your surgical date
5. Not currently pregnant
6. Don't have a history of upper quadrant lymph node dissection, endothelial dysfunction
7. Don't have an active infection or are you currently diagnosed and fighting cancer
8. Don't bruise easily and/or have a bleeding disorder

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
shoulder Isometric strength | 6 weeks
  resisted isometric strength using dynamotor
shoulder Isometric strength | 12 weeks
  resisted isometric strength using dynamotor
shoulder Isometric strength | 6 months
  resisted isometric strength using dynamotor
shoulder function- (CKCUEST) | 6 months
  Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST)
shoulder function- (UQYBT) | 6 months
  Upper Quarter Y Balance Test (UQYBT)
shoulder function-(SSPT) | 6 months
  Seated Shotput Test (SSPT)

SECONDARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 6 weeks
  report self pain rating
Numerical Pain Rating Scale (NPRS) | 12 weeks
  report self pain rating
Numerical Pain Rating Scale (NPRS) | 6 months
  report self pain rating
Shoulder Pain and Disability Index (SPADI) | 6 weeks
  self reported patient outcomes
Shoulder Pain and Disability Index (SPADI) | 12 weeks
  self reported patient outcomes
Shoulder Pain and Disability Index (SPADI) | 6 months
  self reported patient outcomes
Single Assessment Numeric Evaluation (SANE) | 6 weeks,
  self reported patient outcomes
Single Assessment Numeric Evaluation (SANE) | 12 weeks
  self reported patient outcomes
Single Assessment Numeric Evaluation (SANE) | 6 months
  self reported patient outcomes
Quick Disabilities of Arm, Shoulder, Hand (QDASH) | 6 weeks
  self reported patient outcomes
Quick Disabilities of Arm, Shoulder, Hand (QDASH) | 12 weeks
  self reported patient outcomes
Quick Disabilities of Arm, Shoulder, Hand (QDASH) | 6 months
  self reported patient outcomes
ROM | 6 weeks
  shoulder Range of motion using the digital inclinometer
ROM | 12 weeks
  shoulder Range of motion using the digital inclinometer
ROM | 6 months
  shoulder Range of motion using the digital inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- Keller Army Community Hospital - ARVIN, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Following the completion of this study, subject will have the option to allow, or not allow the researchers to keep your data and use it in the future. At the end of the consent form subject will choose to give permission, or not, to use protected health information and study data (non-protected health information) for future research studies. Following study completion, we will remove anything that might identify subject from the information. If subject chooses so, the remaining de-identified information may then be used for future research studies or given to another investigator without getting additional permission from the subject. If we do want to use the information or give the information to another investigator for future research, a review board will decide whether this is allowed.